CLINICAL TRIAL: NCT04981184
Title: Informative of Surface Electromyography and Determination of Prognostic Factors in Assessing the Probability of Recovery of Balance and Gait Parameters in Patients With Ischemic Stroke on Acute Rehabilitation
Brief Title: Informative of Surface Electromyography and Prognostic Factors in Assessing the Recovery of Balance and Gait After Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Ieva Žemaitienė, Ieva Žemaitienė, PT, Lithuanian University of Health Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BE-2-67
Record Dates: First submitted 2021-07-03; First posted 2021-07-28 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Brain Ischemia
Keywords: Surface Electromyography; Gait; Balance; Ischemic stroke
MeSH Terms: conditions — Brain Ischemia; Ischemic Stroke | interventions — Gait

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gait and balance measurement (Other): Gait analysis with surface electromyography measurement: surface electromyography signals (of affected and non-affected legs), gait and stance parameters are collected while the patient walks for 30 seconds on the treadmill with integrated sensor equipment (for measuring the force distribution).
  Balance analysis with Biodex balance system SD: measurements of postural stability, fall risk, limits of stability, sensory integration are collected.
  Interventions: Device: Gait and balance measurement

INTERVENTIONS:
Device: Gait and balance measurement — Virtual gait training procedures are included. Balance training procedures with Biodex Balance system are included too.

SUMMARY:
The aim of the biomedical research is to determine the informativeness and prognostic factors of surface electromyography by assessing the probability of recovery of balance and gait parameters in the second stage of rehabilitation of persons with cerebral infarction.

ELIGIBILITY:
Inclusion Criteria:

* Cerebral infarction for the first time;
* Age from 18 to 89 years old;
* Muscle strength according to the Oxford scale is 3-5 points;
* Able to walk without the help of others;
* Is able to communicate and understand instructions properly;
* Agrees to participate in the study (voluntary, explicit, informed written consent to participate).

Exclusion Criteria:

* Muscle strength according to the Oxford scale is 0-2 points;
* Unable to walk without the help of others;
* Sensorimotor aphasia or other perceptual disorders;
* Do not sign the informed consent.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-07-22 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Muscle strength by Oxford scale | Baseline
  Testing key muscles from the lower extremities (muscle rectus femoris, muscle biceps femoris, muscle gastrocnemius, lateral head, muscle tibialis anterior) against the examiner's resistance and grading the patient's strength on a 0 (No contraction) to 5 (Movement against gravity with full resistance) scale.
Gait analysis with surface electromyography: Load change (seconds) | Baseline, approximately 2 days before the end of acute rehabilitation
  Time change heel to forefoot.
Gait analysis with surface electromyography: Maximum force (Newton) | Baseline, approximately 2 days before the end of acute rehabilitation
  The average maximum force change reached in N/cm² for the three zones: toes, mid-foot and heel.
Gait analysis with surface electromyography: Maximum pressure (Newtons /square centimeter (N/cm²)) | Baseline, approximately 2 days before the end of acute rehabilitation
  The average maximum pressure reached in N/cm² for the three zones: toes, mid-foot and heel (left and right legs separately).
Gait analysis with surface electromyography: Time maximum force (percentage of stance time) | Baseline, approximately 2 days before the end of acute rehabilitation
  The change of the average point in time within a gait cycle where the maximum values for the three zones: toes, mid-foot and heel were collected in Newton.
Gait analysis with surface electromyography: Contact time (percentage of stance time) | Baseline, approximately 2 days before the end of acute rehabilitation
  The average contact time change of the three zone toes, mid-foot and heel as a percentage.
Gait analysis with surface electromyography: Length of the gait line (millimeters) | Baseline, approximately 2 days before the end of acute rehabilitation
  The change from baseline of the progression of the center of pressure of all the steps recorded of one side of the body (left and right side of body separately).
Gait analysis with surface electromyography: Anterior/Posterior Position (millimeters) | Baseline, approximately 2 days before the end of acute rehabilitation
  The shift change forwards or backwards of the Center of pressure.
Gait analysis with surface electromyography: Lateral symmetry (millimeters) | Baseline, approximately 2 days before the end of acute rehabilitation
  The change from baseline of the left /right shift of the center of pressure, taking all the steps into consideration. A negative value indicates a shift to the left, and a positive value, a shift to the right.
Gait analysis with surface electromyography: Step time (seconds) | Baseline, approximately 2 days before the end of acute rehabilitation
  Time change during the phase within a gait cycle between the heel contact of one side of the body and the heel contact of the contralateral side.
Gait analysis with surface electromyography: Cadence (steps/minutes) | Baseline, approximately 2 days before the end of acute rehabilitation
  Change from baseline of step frequency.
Gait analysis with surface electromyography: Velocity (kilometers/hour) | Baseline, approximately 2 days before the end of acute rehabilitation
  Average gait speed change from baseline during the analyzed measuring interval (30 seconds).
Gait analysis with surface electromyography: Stance phase (percentage) | Baseline, approximately 2 days before the end of acute rehabilitation
  The phase of a gait cycle change in which the foot has contact with the ground.
Gait analysis with surface electromyography: Swing phase (percentage) | Baseline, approximately 2 days before the end of acute rehabilitation
  Change from baseline of the phase of a gait cycle during which the foot has no contact with the ground.
Gait analysis with surface electromyography: Double stance phase (percentage) | Baseline, approximately 2 days before the end of acute rehabilitation
  The phase change from baseline during a gait cycle that begins at contralateral initial contact (when the heel of the contralateral side touches the ground) and ends at toe off of the viewed side of the body.
Gait analysis with surface electromyography: Foot rotation (degree) | Baseline, approximately 2 days before the end of acute rehabilitation
  The change from baseline of the angle between the longitudinal axis of the foot and the walking direction.
Gait analysis with surface electromyography: Step length (centimeters) | Baseline, approximately 2 days before the end of acute rehabilitation
  Change of the distance between the heel contact of one side of the body and the heel contact of the contralateral side.
Gait analysis with surface electromyography: Stride length (centimeters) | Baseline, approximately 2 days before the end of acute rehabilitation
  the distance change between two heel contacts on the same side of the body.
Gait analysis with surface electromyography: Step width (centimeters) | Baseline, approximately 2 days before the end of acute rehabilitation
  The distance change between the right and left foot.
Gait analysis with surface electromyography: surface electromyography signals (microvolts) | Baseline, approximately 2 days before the end of acute rehabilitation
  Surface electromyography measurements of key muscles (muscle rectus femoris, muscle biceps femoris, muscle gastrocnemius, lateral head, muscle tibialis anterior) with a disposable dual surface electrode. Change of surface electromyography signals during walking on treadmill for 30 seconds.
Stance analysis: Step width (centimeters) | Baseline, approximately 2 days before the end of acute rehabilitation
  Change from baseline of the averaged load distribution of the left and right forefoot or heel, as well as the load distribution of the left and right contact surface in per cent.

SECONDARY OUTCOMES:
Biodex Balance System (BBS): Postural Stability Test (Overall stability index) | Baseline, approximately 2 days before the end of acute rehabilitation
  The BBS will be used to assess postural performance of participants. The movable platform of the BBS allows up to 20° of surface tilt in anterior-posterior and medial-lateral directions. The device is equipped with computer software (Biodex, version 3.1; Biodex Medical Systems). Platform Setting 8. Test Trial Time 20 secs. A high number is indicative of a lot of motion, which is indicative of the patient having trouble balancing. Change from baseline postural stability by overall stability index.
Biodex Balance System (BBS): Limits of Stability Test (seconds) | Baseline, approximately 2 days before the end of acute rehabilitation
  During test, patients must shift their weight to move the cursor from the center target to a blinking target and back as quickly and with as little deviation as possible. Platform Setting STATIC. Direction control - OVERALL. Faster - better. Time change of limit of stability test.
Biodex Balance System (BBS): Limits of Stability Test (score) | Baseline, approximately 2 days before the end of acute rehabilitation
  During test, patients must shift their weight to move the cursor from the center target to a blinking target and back as quickly and with as little deviation as possible. Platform Setting STATIC. Direction control - OVERALL. The goal - 65 scores and more. Score change of limit of stability test.
Biodex Balance System (BBS): A fall risk test (scores) | Baseline, approximately 2 days before the end of acute rehabilitation
  Test results are compared to age dependent normative data. Scores higher than normative values suggest further assessment. Platform Setting 12-8. Test Trial Time 20 seconds. Direction control - OVERALL. Patient's aged 54-71 years' normative scores are 0.9-3.7 scores, 72-89 years' normative scores are 2-4 scores, 36-53 years' normative scores are 0.7-3.1 scores, 17-35 years' normative scores are 0.7-2.1 scores. Change from baseline a fall risk by scores.
Biodex Balance System (BBS): Clinical Test of Sensory Integration of Balance(CTSIB) (sway index) | Baseline, approximately 2 days before the end of acute rehabilitation
  The test assesses how well a patient can integrate sensory information to maintain balance. Change from baseline the CTSIB test by the patient's sway index, which represents the mean absolute deviation of the patient's average position during a test. The higher the sway index, the more unsteady the person was during the test. Test Trial Time 30 seconds. The test performs with the patient standing on a firm and foam platform with the eyes open and closed. Measure Sway index of Composite Score.
Biodex Balance System (BBS): Balance Error Scoring System (sway index) | Baseline, approximately 2 days before the end of acute rehabilitation
  A test consists of three positions (Double Leg Stance, Single Leg Stance and Tandem Leg Stance) on two types of platforms (firm and foam) for a total of six conditions. With the Balance System SD, time and error counting is replaced with a measure of sway. Change from baseline balancing errors by Sway index of Composite Score. The higher the sway index, the more unsteady the person was during the test. Test Trial Time 20 seconds

CONTACTS AND LOCATIONS:
Overall Officials: Eglė Lendraitienė, PhD, Principal Investigator — LUHS
Locations (1):
- LUHS hospital Kaunas Clinics Rehabilitation hospital of Kulautuva, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: No